CLINICAL TRIAL: NCT05335720
Title: Study to Evaluate the Efficacy and Safety of EASYEF® in Acute Wound (Split-thickness Skin Graft Donor Site)
Brief Title: Efficacy and Safety Evaluation of EASYEF® in Acute Wound (Split-thickness Skin Graft Donor Site)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT. Daewoong Infion (Industry)
Collaborators: Equilab International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_EGFCS
Record Dates: First submitted 2022-04-06; First posted 2022-04-19 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Skin Graft Scar; Split-Thickness Skin Graft (STSG)
Keywords: EGF; Epidermal Growth Factor; rhEGF; recombinant human Epidermal Growth Factor; Acute wound; Skin graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): 1. EASYEF® + moist gauze EASYEF® is applied directly on the wound surface then moist dressing is used as primary dressing before covered with dry gauze. All dressings are fixed with elastic bandage.
  2. Tulle gauze + moist gauze Tulle gauze is applied directly on the wound surface then moist dressing is used as primary dressing before covered with dry gauze. All dressings are fixed with elastic bandage.
  Interventions: Drug: rhEGF
- Cohort 2 (Active Comparator): 1. EASYEF® + tulle gauze + moist gauze EASYEF® is applied directly on the wound surface then tulle gauze and moist gauze is used as primary dressing before covered with dry gauze. All dressings are fixed with elastic bandage.
  2. Tulle gauze + moist gauze Tulle gauze is applied directly on the wound surface then moist dressing is used as primary dressing before covered with dry gauze. All dressings are fixed with elastic bandage.
  Interventions: Drug: rhEGF

INTERVENTIONS:
Drug: rhEGF — EASYEF® spray 50 mcg, sprayed twice a day for 14 days.
  Other Names: EASYEF®

SUMMARY:
This study is a prospective study, randomized, using control, open-label, single-center to evaluate the efficacy and safety of EASYEF® in acute wound (split-thickness skin graft donor site). A total of 10 subjects are randomly allocated. Subjects who meet the final inclusion and exclusion criteria are randomized to the test cohorts in a ratio of 1:1:1.

DETAILED DESCRIPTION:
This study was intended to determine the effect of EGF on acute wounds such as trauma, surgical wounds and burns. But in this study, skin graft donor site wounds were used because they were the most representative for acute wounds and the depth and extent of the wounds could be controlled. EGF is known pharmacologically to accelerate epithelial cell proliferation, fibroblast cells and endothelial cells. Giving EGF in acute wounds is expected to accelerate wound healing and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have donor wounds on the vertical (upper and lower) lines of the thigh through skin grafted surgery due to trauma, ulcers, burns, and incisional surgical defects.
* The size of the donor follows the standard and the distance between the two skin transplants is at least 2 cm.
* Patients who are expected to be able to successfully complete or benefit from this examination are based on appropriate medical assessment.
* Patients is willing to be treated 7 days as inpatient and treated as outpatient for maximum 7 days with homecare nurse visit.
* Patients is willing to stay near the hospital and visit the hospital after the donor site wound is declared healed by doctor.
* Patients who decided and agreed in writing to enroll in this study at their own will.
* Patients aged 18 and up

Exclusion Criteria:

* Patients with different skin donor site can influence the results of the study.
* Patients who have other diseases that can interfere with wound healing such as immunosuppressive, metabolic collagen, peripheral vascular obstructive disease (PAOD), systemic vasculitis, and others.
* Patients have the talent for keloid formation.
* Patients have uncontrolled diabetes and diabetes with complications.
* Patients with liver disease, kidney disease, and other serious diseases that can affect this study.
* Patients who are deemed difficult to carry out the study by the investigators.
* Women who are pregnant, lactation or not using reliable methods of contraception and who do not consent to continue contraception for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the wound healing time of each skin graft donor site | 14 days
  The definition of 'wound healing' is when there is no more exudate in the skin graft donor and the skin is covered with epithelial tissue in a milky light pink color and there is no pain. Healing time (morning or afternoon) evaluation and pain scale (11-point NRS (Numeric Rating Scale); 0 = No pain, 5 = Moderate pain, and 10 = Worst possible pain) will be assessed.

SECONDARY OUTCOMES:
Adverse Events | 14 days
  In order to confirm the adverse events (AE), it is confirmed through the questionnaire of investigators and the physical examination. If an adverse event occurs, record the timing of the adverse event, the duration, the extent of the adverse event, and the causal relationship.
Photograph evaluation | 14 days
  During the change of dressing in the morning and evening, photograph was taken to evaluate the re-epithelization improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- RSPAD Gatot Soebroto, Central Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided